CLINICAL TRIAL: NCT00435292
Title: A Double-Blind, Randomized, Placebo Controlled, Parallel Group, Multi Center Study of Flavocoxid ( Limbrel) vs Naproxen in Subjects With Moderate-Severe Osteoarthritis of the Knee
Brief Title: Study of Flavocoxid (Limbrel) vs Naproxen in Subjects With Mod-Severe Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LOA-03P
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2008-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Naproxen; flavocoxid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- flavocoxid 250 mg (Experimental): flavonoid mixture
  Interventions: Dietary Supplement: flavocoxid 250 mg
- flavocoxid 500 mg (Active Comparator): flavonoid mixture
  Interventions: Dietary Supplement: flavocoxid 500 mg
- naproxen (Active Comparator): nonsteroidal antiinflammatory drug
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Naproxen — nonsteroidal anti-inflammatory drug
  Other Names: naprosyn
  Arms: naproxen
Dietary Supplement: flavocoxid 250 mg — flavonoid mixture
  Other Names: Limbrel 250 mg
  Arms: flavocoxid 250 mg
Dietary Supplement: flavocoxid 500 mg — flavonoid mixture
  Other Names: limbrel 500 mg
  Arms: flavocoxid 500 mg

SUMMARY:
Randomized, double-blind, placebo controlled parallel group, multi center study in subjects with moderate-severe osteoarthritis.

DETAILED DESCRIPTION:
This will be a randomized, double blind, placebo controlled, parallel group, multi-center study in subjects with moderate-severe OA. Subjects will be randomized to receive flavocoxid 250 mg bid, flavocoxid 500 mg bid, naproxen 500 mg bid or placebo in a 2:2:2:1 ratio. Subjects will take study materials twice daily for twelve (12) weeks. After the 12 week visit subjects in the placebo arm will be re-randomized to the two flavocoxid arms. All subjects will then continue on the study for an additional 12 weeks.

Subjects will keep a diary noting date of onset of symptom change (better or worse), adverse events and cost of all aspects of medical care related directly or indirectly to osteoarthritis.

Laboratory studies for inflammatory markers will be drawn and archived at baseline and at the 12 week visit. In addition, a subgroup of subjects will have arthrocenteses performed at baseline and the 12 week visit and the synovial fluid archived for study of intra-articular inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* OA of the Knee
* K-L Grade 2-3
* Positive response to NSAIDS

Exclusion Criteria:

* K-L grade 1 0r 4 OA of the knee
* History of GI Bleed within past 5 years
* Chronic bleeding disorder

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2006-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Levy, MD, Study Director — Primus Pharmaceuticals,Inc; Alan Kivitz, MD, Principal Investigator — Private Practice
Locations (1):
- Primus Pharmaceuticals, Inc, Scottsdale, Arizona, United States